CLINICAL TRIAL: NCT03828994
Title: Technology Based Community Health Nursing(TECH-N) to Prevent Recurrent STIs After PID
Brief Title: Technology Based Community Health Nursing(TECH-N) to Prevent Recurrent STIs After PID II
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NA_00068846-2; R01NR013507-03 (NIH)
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Inflammatory Disease
Keywords: Pelvic Inflammatory Disease(PID); Community Health Nursing; Adolescents; Text Messaging; mobile health (mhealth)
MeSH Terms: conditions — Pelvic Inflammatory Disease

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TECH-PN (Experimental): Participants receive community health nurse visits, text-messaging support, additional testing and field based visits with a nurse practitioner.
  Interventions: Behavioral: Tech-PN
- TECH-N (No Intervention): Participants receive enhanced standard of care with community health nurse visits and text-messaging support.

INTERVENTIONS:
Behavioral: Tech-PN — * text messaging(daily medication reminders and tri-weekly messages following the 14-day treatment period)
  * enhanced community health nurse visits on day 3-5, 14 and 30
  * field based treatment visits
  * clinical assistance with notification, testing and treatment
  Arms: TECH-PN

SUMMARY:
The investigators are enrolling 150 young women 13-25 years old diagnosed with pelvic inflammatory disease (PID) in Baltimore to receive community health nurse (CHN) clinical support visits and short messaging system communication support for 30 days. The investigators' intervention group(TECH-PN) will receive additional testing and treatment in the field. The investigators hypothesize that repackaging the recommended Centers for Disease Control and Prevention (CDC) follow-up visit using a technology-enhanced community health nursing intervention (TECH-N) with integration of an evidence-based sexually transmitted infection (STI) prevention curriculum will reduce rates of short-term repeat infection by improving adherence to PID treatment and reducing unprotected intercourse and be more cost-effective compared with outpatient standard of care (and hospitalization).

DETAILED DESCRIPTION:
Pelvic Inflammatory Disease (PID) is a common, serious reproductive disorder that is associated with significant adverse reproductive health outcomes such as ectopic pregnancy, tubal infertility, chronic pelvic pain, and significant reductions in health-related quality of life for affected patients. The Technology Enhanced Community Health (TECH) Nursing Study has further demonstrated that the biological milieu associated with PID is more complicated than the Centers for Disease Control and Prevention (CDC) treatment guidance indicates, leaving women without adequate treatment for Mycoplasma genitalium (MG) and Trichomonas vaginalis (TV). The broad-spectrum antibiotics recommended by the CDC for syndromic PID management are suboptimal because: 1) MG is often resistant to doxycycline (standard therapy) and macrolides such as Azithromycin (alternative therapy) and 2) metronidazole (effective for TV) is an optional add-on to standard PID treatment that is inconsistently prescribed at diagnosis. Further MG was not officially considered in CDC STI treatment guidelines until release until 2015, testing is only available in large research laboratories, and the paucity of data from randomized trials limits the scope of the CDC's recommendations. Finally, while there are no public health control programs in the United States for MG and TV, recurrent and persistent infection with MG and TV is associated with ongoing inflammation in the female genital tract and increased risk for secondary STI and HIV infection due to unhealthy shifts in vagina microbiota. The goals of this study are to leverage novel STI diagnostics (new MG macrolide resistance testing and TV testing) with the investigators' demonstrated ability to reach vulnerable youth to treat adolescents and young adult women with mild-moderate PID with precision based on the actual diagnoses rather than suboptimal syndromic management. The investigators will add genomic analysis of vaginal specimens to assess compositional changes in the five vaginal Lactobacilli community state types associated with optimal vaginal health to determine if TECH-precision-nursing (TECH-PN) protocols for field treatment tailored to STI results reduces the inflammatory response observed with active vaginal infections. The investigators hypothesize that by further repackaging the investigators' previous successful TECH-N intervention protocol and translating bench science into precision healthcare, the investigators will further reduce the risk of recurrent infection, potentially restore vaginal health for PID- affected patients, and add new knowledge that advances public health control of STIs and has the potential to reduce the observed STI disparities after PID in urban youth.

ELIGIBILITY:
Inclusion Criteria:

* Mild-moderate PID
* Outpatient treatment disposition
* Permanently reside in the Baltimore Metropolitan area
* Willing to sign informed consent & be randomized

Exclusion Criteria:

* Pregnant
* Concurrent diagnosis of Sexual Assault
* Unable to communicate/complete study procedures

Ages: 13 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-02-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Rate of STI Trichomonas vaginalis | 3 months
  Trichomonas infection assessed with Aptima vaginal swab, tested using the Gen-Probe transcription mediated amplification (TMA) research assay.
Rate of STI Mycoplasma genitalium | 3 months
  Mycoplasma infection assessed with Aptima vaginal swab, tested using the Gen-Probe transcription mediated amplification (TMA) research assay.
Vaginal health as assessed by proportion of high Lactobacilli community state-type 1 properties (CST) | 90 days
  Vaginal microbiota will be identified with a 16S ribosomal RNA (16S rRNA) amplicon sequencing analysis. The proportion of rRNA assigned to the bacterial genera Lactobacillus will be measured for each sample. CST (I, II, II, IV) will be assigned based on taxa identified.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Trent, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anders J, Hill A, Chung SE, Butz A, Rothman R, Gaydos C, Perin J, Trent M. Patient Satisfaction and Treatment Adherence for Urban Adolescents and Young Adults with Pelvic Inflammatory Disease. Trauma Emerg Care. 2018 Jan;3(1):10.15761/TEC.1000152. doi: 10.15761/TEC.1000152. Epub 2017 Aug 25. PMID 29756068
- [Background] Trent M, Chung SE, Gaydos C, Frick KD, Anders J, Huettner S, Rothman R, Butz A. Recruitment of Minority Adolescents and Young Adults into Randomised Clinical Trials: Testing the Design of the Technology Enhanced Community Health Nursing (TECH-N) Pelvic Inflammatory Disease Trial. Eur Med J Reprod Health. 2016 Aug;2(1):41-51. PMID 27617108
- [Background] Butz AM, Gaydos C, Chung SE, Johnson BH, Huettner S, Trent M. Care-Seeking Behavior After Notification Among Young Women With Recurrent Sexually Transmitted Infections After Pelvic Inflammatory Disease. Clin Pediatr (Phila). 2016 Oct;55(12):1107-12. doi: 10.1177/0009922816662863. Epub 2016 Aug 8. PMID 27507807
- [Background] Munoz Buchanan CR, Chung SE, Butz A, Perin J, Gaydos C, Trent M. Perceived Social Support, Parental Notification, and Parental Engagement after Pelvic Inflammatory Disease among Urban Adolescent and Young Adults. Pediatr Neonatal Nurs. 2016;4(1):12-16. doi: 10.17140/pnnoj-4-124. Epub 2016 Nov 17. PMID 28280783
- [Background] Tabacco L, Chung SE, Perin J, Huettner S, Butz A, Trent M. Relationship Status and Sexual Behaviors in Post-Pelvic Inflammatory Disease (PID) Affected Urban Young Women: A Sub-Study of a Randomized Controlled Trial. Int Arch Nurs Health Care. 2018;4(1):088. doi: 10.23937/2469-5823/1510088. Epub 2018 Jan 10. PMID 30221216
- [Background] Haggerty CL, Totten PA, Tang G, Astete SG, Ferris MJ, Norori J, Bass DC, Martin DH, Taylor BD, Ness RB. Identification of novel microbes associated with pelvic inflammatory disease and infertility. Sex Transm Infect. 2016 Sep;92(6):441-6. doi: 10.1136/sextrans-2015-052285. Epub 2016 Jan 29. PMID 26825087
- [Background] Mitchell CM, Haick A, Nkwopara E, Garcia R, Rendi M, Agnew K, Fredricks DN, Eschenbach D. Colonization of the upper genital tract by vaginal bacterial species in nonpregnant women. Am J Obstet Gynecol. 2015 May;212(5):611.e1-9. doi: 10.1016/j.ajog.2014.11.043. Epub 2014 Dec 16. PMID 25524398
- [Background] Molenaar MC, Singer M, Ouburg S. The two-sided role of the vaginal microbiome in Chlamydia trachomatis and Mycoplasma genitalium pathogenesis. J Reprod Immunol. 2018 Nov;130:11-17. doi: 10.1016/j.jri.2018.08.006. Epub 2018 Aug 22. PMID 30149363
- [Background] Wang Y, Zhang Y, Zhang Q, Chen H, Feng Y. Characterization of pelvic and cervical microbiotas from patients with pelvic inflammatory disease. J Med Microbiol. 2018 Oct;67(10):1519-1526. doi: 10.1099/jmm.0.000821. Epub 2018 Aug 16. PMID 30113305
- [Result] Zheng X, O'Connell CM, Zhong W, Poston TB, Wiesenfeld HC, Hillier SL, Trent M, Gaydos C, Tseng G, Taylor BD, Darville T. Gene Expression Signatures Can Aid Diagnosis of Sexually Transmitted Infection-Induced Endometritis in Women. Front Cell Infect Microbiol. 2018 Sep 20;8:307. doi: 10.3389/fcimb.2018.00307. eCollection 2018. PMID 30294592
- [Derived] Perin J, Anders J, Barfield A, Gaydos C, Rothman R, Matson PA, Huettner S, Toppins J, Trent M. Undermining the Translational Potential of Clinical Research With Adolescents and Young Adults: Differential Enrollment in Randomized Clinical Trials During COVID-19. Sex Transm Dis. 2024 Oct 1;51(10):681-685. doi: 10.1097/OLQ.0000000000001994. Epub 2024 May 1. PMID 38691409
- [Derived] Trent M, Perin J, Rowell J, Shah M, Anders J, Matson P, Brotman RM, Ravel J, Sharps P, Rothman R, Yusuf HE, Gaydos CA. Using Innovation to Address Adolescent and Young Adult Health Disparities in Pelvic Inflammatory Disease: Design of the Technology Enhanced Community Health Precision Nursing (TECH-PN) Trial. J Infect Dis. 2021 Aug 16;224(12 Suppl 2):S145-S151. doi: 10.1093/infdis/jiab157. PMID 34396402